CLINICAL TRIAL: NCT00853593
Title: Model 4396 Left Ventricular Lead Study
Brief Title: Model 4396 Left Ventricular (LV) Lead Study
Acronym: 4396
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2011-12-05 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac pacing; cardiac resynchronization therapy; left ventricular lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Model 4396 LV Lead (Experimental): Non-randomized study.
  Interventions: Device: Pacing Lead

INTERVENTIONS:
Device: Pacing Lead — implant and follow-up of study device

SUMMARY:
This study is designed to show that a new lead, which paces the left bottom chamber (left ventricle) of the heart, is safe and effective. Using a lead on the left side of the heart has been shown to potentially improve heart failure symptoms. The shape and size of this new lead may make it a good choice for patients or physicians.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, non-randomized design. All consented patients who meet all inclusion and no exclusion criteria may receive the investigational lead. The study design has statistical power to show safety at one-month after implant. It also has statistical power to show effectiveness at one-month and three-months after implant.

ELIGIBILITY:
Inclusion Criteria:

* CRT/Cardiac Resynchronization Therapy-Defibrillator (CRT-D) indications, New York Heart Association (NYHA) III and IV, indicated for implantable cardiac defibrillator (ICD) if CRT-D is implanted, patient consent, geographically stable

Exclusion Criteria:

* LV lead implant attempt in last 30 days, unstable angina or acute myocardial infarction (MI) in past 30 days, coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) in past 3 months, contraindicated for transvenous pacing, heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Exner, MD, Principal Investigator — Foothills Hospital (University of Calgary); Daniel Gras, MD, Principal Investigator — Nouvelles Cliniques Nantaises
Locations (31):
- United States (19):
  - Pasadena, California
  - Sacramento, California
  - Atlantis, Florida
  - Atlanta, Georgia
  - Hinsdale, Illinois
  - Davenport, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Saint Louis Park, Minnesota
  - Saint Paul, Minnesota
  - Liverpool, New York
  - New York, New York
  - Durham, North Carolina
  - Portland, Oregon
  - York, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Morgantown, West Virginia
- Bendigo, Australia
- Linz, Austria
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Newmarket, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Aarhus, Denmark
- France (2):
  - Nantes
  - Toulouse
- Treviso, Italy
- Riyadh, Saudi Arabia

RESULTS

PARTICIPANT FLOW:
Groups:
- Model 4396 LV Lead: Subjects successfully implanted with a Model 4396 LV lead.
Period: Overall Study
Arm/Group | Model 4396 LV Lead
Started | 197
Implant Attempted | 193
Model 4396 Lead Attempted | 164
Completed | 152
Not Completed | 45
Not completed — Subjects did not receive a 4396 lead | 12
Not completed — Model 4396 lead not attempted | 29
Not completed — Implant not attempted | 4

BASELINE CHARACTERISTICS:
Groups:
- Model 4396 LV Lead: Subjects underwent Model 4396 left ventricular lead implant attempt
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 193
Age, Categorical [Count of Participants; unit: Participants] — All subjects who underwent an implant attempt (193) were included in the study population analysis.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 62
    >=65 years | 131
Age, Continuous [Mean (Standard Deviation); unit: years] — All subjects who underwent an implant attempt (193) were included in the study population analysis.
  years | 69.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants] — All subjects who underwent an implant attempt (193) were included in the study population analysis.
  Participants
    Female | 53
    Male | 140
Region of Enrollment [Number; unit: participants] — All subjects who underwent an implant attempt (193) were included in the study population analysis.
  participants
    France | 10
    United States | 125
    Canada | 47
    Australia | 2
    Denmark | 3
    Austria | 6
New York Heart Association [Number; unit: participants] — All subjects who underwent an implant attempt (193) were included in the study population analysis
  participants
    Class III | 192
    Class IV | 1
Race/Ethnicity [Number; unit: participants] — All subjects who underwent an implant attempt (193) were included in the study population.
  participants
    Asian | 2
    Black or African American | 9
    Hispanic or Latino | 6
    Native Hawaiian or Pacific Islander | 1
    White/Caucasian | 168
    Subject chose not to provide information | 6
    Other | 1
Intrinsic QRS Width [Mean (Standard Deviation); unit: Milliseconds] — All subjects who underwent an implant attempt (193) were included in the study population analysis.
  Milliseconds | 154.1 (24.9)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: Percent] — All subjects who underwent an implant attempt (193) were included in the study population analysis. Note, one subject did not have a LVEF within 365 days of baseline and a study deviation was reported for not meeting inclusion/exclusion criteria.
  Percent | 25.7 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Safety (Subjects Without a Model 4396 Lead Related Complication)
Description: A subject who was free of a Model 4396 lead related complication by the one month visit. All adverse events (AE) in the time frame were recorded at the subject's center and assessed by a centralized Adverse Event Advisory Committee (AEAC). The AEAC determined whether an AE was a complication and whether the event was related to the Model 4396 lead. A complication is an AE that results in death, termination of significant device function or invasive intervention (any therapy that penetrates the skin including administration of intramuscular (IM) and parenteral (IV) fluids).
Time Frame: One month
Population: Subjects who underwent a Model 4396 left ventricular (LV) lead implant attempt and had a 1 month follow-up visit.
Measure: Number; unit: participants
Groups:
- Model 4396 LV Lead: Subjects who underwent a Model 4396 left ventricular lead implant attempt
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 163
participants | 155 [90.6 to 95]
Statistical Analysis 1: Comparison: Model 4396 LV Lead; Test type: Superiority or Other; One sample proportion = .951, 95% CI 1-sided [lower limit .906] — The Model 4396 lead will be considered safe if the proportion of subjects free of Model 4396 lead-related complications at one month post-implant is greater than 80% (i.e. the one sided 95% lower confidence bound must be at least 80%)

2. Primary Outcome: Efficacy: Distal Tip Electrode Voltage Threshold
Description: Subjects' distal tip electrode voltage threshold was collected at the one month visit. The Model 4396 was considered effective if the mean voltage threshold was less than 3.0 Volts. Voltage threshold was collected using LV tip to Right Ventricular (RV) coil configuration at 0.5 milliseconds [ms]. Voltage threshold is the minimum energy required from the device to consistently pace the ventricle.
Time Frame: One month
Population: Only subjects with pacing thresholds captured at 0.5 ms were included in the analysis.
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Model 4396 LV Lead: Subjects with tip electrode capture at 0.5ms at 1-month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 139
Volts | 1.6 (1.4)
Statistical Analysis 1: Comparison: Model 4396 LV Lead; Test type: Superiority or Other; One sample mean = 1.6, 95% CI 1-sided [upper limit 1.8], Standard Deviation 1.4

3. Primary Outcome: Efficacy: Proximal Ring Voltage Threshold
Description: Subject's proximal ring electrode voltage threshold was collected at the three months visit. The Model 4396 was considered effective if the mean voltage threshold was less than 3.0 Volts.
Time Frame: Three months
Population: Subjects with ring electrode threshold captured at 0.5 ms at 3-month
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Model 4396 LV Lead: Subjects with ring electrode threshold captured at 0.5ms at 3-month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 121
Volts | 2.3 (2.0)
Statistical Analysis 1: Comparison: Model 4396 LV Lead; Test type: Superiority or Other; One sample mean = 2.3, 97.5% CI 1-sided [upper limit 2.7], Standard Deviation 2.0

4. Secondary Outcome: Subjects Successfully Implanted With Model 4396 Lead
Description: A successful implant occurs when the Model 4396 lead is implanted in a left ventricular vein and functions appropriately. A Model 4396 implant attempt was defined as any time when a Model 4396 lead was introduced into the body.
Time Frame: During implant procedure.
Population: Subjects who underwent Model 4396 LV implant attempt.
Measure: Number; unit: participants
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 164
participants | 152
Statistical Analysis 1: Comparison: Model 4396 LV Lead; Test type: Superiority or Other; One sample proportion = .927, 95% CI 2-sided [.887 to .967]

5. Secondary Outcome: Subjects Successfully Implanted With Any Transvenous LV Lead After Cannulation
Description: A successful implant after cannulation occurs when the coronary sinus (CS) is successfully cannulated and a left ventricular lead (any transvenous LV lead) is implanted in a left ventricular vein and functions appropriately. An implant attempt of any transvenous LV lead was defined as any time when a transvenous LV lead was introduced into the body.
Time Frame: During implant procedure.
Population: Subjects with successful CS cannulation after an implant attempt.
Measure: Number; unit: participants
Groups:
- Any Transvenous LV Lead: Subjects who underwent an implant attempt with successful CS cannulation.
Arm/Group | Any Transvenous LV Lead
Number analyzed (Participants) | 191
participants | 185
Statistical Analysis 1: Comparison: Any Transvenous LV Lead; Test type: Superiority or Other; One sample proportion = .969, 95% CI 2-sided [.944 to .993]

6. Secondary Outcome: Subjects Successfully Implanted With Any Transvenous LV Lead
Description: A successful implant occurs when any transvenous LV lead is implanted in a left ventricular vein functions appropriately.
Time Frame: During implant procedure.
Population: Subjects who underwent an implant attempt.
Measure: Number; unit: participants
Groups:
- Any Transvenous LV Lead: Subjects who underwent an implant attempt.
Arm/Group | Any Transvenous LV Lead
Number analyzed (Participants) | 193
participants | 185
Statistical Analysis 1: Comparison: Any Transvenous LV Lead; Test type: Superiority or Other; One sample proportion = .959, 95% CI 2-sided [.930 to .987]

7. Secondary Outcome: Subjects Successfully Implanted With Any Medtronic Attain Family LV Lead
Description: A successful implant occurs when any Medtronic Attain Family LV Lead is implanted in a left ventricular vein and functions appropriately. The Attain Family leads include the following models: 4193, 4194, 4195, 4196, and 4396.
Time Frame: During implant procedure.
Population: Subjects who underwent an implant attempt.
Measure: Number; unit: participants
Groups:
- Any Medtronic LV Lead (Attain Family Lead): Subjects who underwent an implant attempt.
Arm/Group | Any Medtronic LV Lead (Attain Family Lead)
Number analyzed (Participants) | 193
participants | 183
Statistical Analysis 1: Comparison: Any Medtronic LV Lead (Attain Family Lead); Test type: Superiority or Other; One sample proportion = .948, 95% CI 2-sided [.917 to .979]

8. Secondary Outcome: Cannulation Time
Description: Cannulation time was defined as the time from insertion of the first coronary sinus (CS) cannulation catheter to the first successful CS cannulation.
Time Frame: During implant procedure.
Population: Subjects successfully implanted with a Model 4396 lead.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 152
minutes | 6.1 (9.0)

9. Secondary Outcome: Fluoroscopy Time
Description: The total time the fluoroscope was imaging (not including biplane fluoroscopy time).
Time Frame: During implant procedure.
Population: Subjects successfully implanted with a Model 4396 lead. Note that one subject's standard fluoroscopy time was not collected and a study deviation was reported.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 151
minutes | 20.6 (13.6)

10. Secondary Outcome: Model 4396 Lead Placement Time
Description: Model 4396 lead placement time was defined as the time from insertion of the successfully implanted lead to the time when it was placed in the first acceptable pacing location.
Time Frame: During implant procedure.
Population: Subjects successfully implanted with a Model 4396 lead. Note that one subject's LV Lead placement time was permanently missing and a study deviation was reported.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 151
minutes | 13.9 (16.3)

11. Secondary Outcome: Total Operation Time
Description: Total operation time was defined as time from initial incision to final closure.
Time Frame: During implant procedure.
Population: Subjects successfully implanted with a Model 4396 lead.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 152
minutes | 97.4 (41.3)

12. Secondary Outcome: Assessment of Lead Handling Characteristics Reported as Acceptable
Description: Implant lead handling characteristics were qualitatively assessed through physician feedback on the Implant Case Report Form (CRF). Physicians were asked for their overall assessment of the lead and results were categorized as acceptable or unacceptable. The number of acceptable responses are summarized.
Time Frame: During implant procedure.
Population: Subjects who underwent a Model 4396 left ventricular lead implant attempt.
Measure: Number; unit: participants
Groups:
- Model 4396 LV Lead: Model 4396 lead implant attempts.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 164
participants | 162

13. Secondary Outcome: Efficacy: Bipolar Voltage Threshold
Description: Subjects' voltage threshold in the bipolar configuration was collected at the one month visit. The Model 4396 was considered effective if the mean voltage threshold (at 0.5 milliseconds [ms]) is less than or equal to 4.0 Volts.
Time Frame: 1 month
Population: Subjects that were implanted with a Model 4396 lead and completed the 1 month visit
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Model 4396 LV Lead: Subjects successfully implanted with a Model 4396 LV lead and completed 1 month visit.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 136
Volts | 2.4 (1.9)
Statistical Analysis 1: Comparison: Model 4396 LV Lead; Test type: Superiority or Other; One sample mean = 2.4, 95% CI 1-sided [upper limit 2.7], Standard Deviation 1.9

14. Secondary Outcome: Characterize Model 4396 Electrical Performance- Tip Electrode: Voltage Threshold
Description: Tip electrode voltage threshold at 0.5 ms was collected at implant, pre-hospital discharge and all scheduled follow-up visits. Voltage threshold values at the 6 month visit are summarized.
Time Frame: 6 month
Population: Subjects with tip electrode threshold captured at 0.5 ms at 6 month
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Model 4396 LV Lead: Subjects with tip electrode threshold captured at 0.5ms at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 128
Volts | 1.5 (1.3)

15. Secondary Outcome: Characterize Model 4396 Electrical Performance- Tip Electrode: Pacing Impedance
Description: Subjects' tip electrode pacing impedance (a measure of electrical resistance) was measured at implant, pre-hospital discharge and all scheduled follow-up visits. Pacing impedance at the 6 month visit is presented here.
Time Frame: 6 month
Population: Subjects with tip electrode pacing impedance at 6 month
Measure: Mean (Standard Deviation); unit: Ohms
Groups:
- Model 4396 LV Lead: Subjects with tip electrode pacing impedance at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 135
Ohms | 571.2 (155.0)

16. Secondary Outcome: Characterize Model 4396 Electrical Performance- Tip Electrode: Sensing
Description: Tip electrode sensing, measured by R-wave amplitude, for the Model 4396 was collected at implant, pre-hospital discharge and all scheduled follow-up visits. Measurements at the 6 month visit are presented here. Sensing is the minimum energy produced by the left ventricle of the heart that the device can sense.
Time Frame: 6 month
Population: Subjects with tip electrode R-wave amplitude at 6 month
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Model 4396 LV Lead: Subjects with ring electrode R-wave amplitude at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 140
mV | 18.3 (6.4)

17. Secondary Outcome: Characterize Model 4396 Electrical Performance- Ring Electrode: Voltage Threshold
Description: Ring electrode voltage threshold at 0.5 ms was collected at implant, pre-hospital discharge and all scheduled follow-up visits. Voltage threshold at the 6 month visit is presented here.
Time Frame: 6 month
Population: Subjects with ring electrode threshold captured at 0.5 ms at 6 month
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Model 4396 LV Lead: Subjects with ring electrode threshold captured at 0.5 ms at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 121
Volts | 2.2 (2.0)

18. Secondary Outcome: Characterize Model 4396 Electrical Performance- Ring Electrode: Pacing Impedance
Description: Subjects' ring electrode pacing impedance was measured at implant, pre-hospital discharge and all scheduled follow-up visits. Pacing impedance at the 6 month visit is presented here.
Time Frame: 6 month
Population: Subjects with ring electrode pacing impedance at 6 month
Measure: Mean (Standard Deviation); unit: Ohms
Groups:
- Model 4396 LV Lead: Subjects with ring electrode pacing impedance at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 134
Ohms | 544.8 (149.2)

19. Secondary Outcome: Characterize Model 4396 Electrical Performance- Ring Electrode: Sensing
Description: Ring electrode sensing, measured by R-wave amplitude, for the Model 4396 was collected only at the implant procedure because the devices allowed in this study are not programmable to collect sensing measurements using the ring electrode. The analyzer was used to collect measurements.
Time Frame: During implant procedure.
Population: Subjects with ring electrode R-wave amplitude at implant
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Model 4396 LV Lead: Subjects with ring electrode R-wave amplitude at implant.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 140
mV | 17.6 (6.6)

20. Secondary Outcome: Characterize Model 4396 Electrical Performance- Bipolar Configuration: Voltage Threshold
Description: Bipolar voltage threshold at 0.5 ms was collected at implant, pre-hospital discharge and all scheduled follow-up visits. Voltage threshold at the 6 month visit is reported here.
Time Frame: 6 month
Population: Subjects with bipolar configuration threshold captured at 0.5 ms at 6 month
Measure: Mean (Standard Deviation); unit: Volts
Groups:
- Model 4396 LV Lead: Subjects with bipolar configuration threshold captured at 0.5ms at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 128
Volts | 2.4 (2.0)

21. Secondary Outcome: Characterize Model 4396 Electrical Performance- Bipolar Configuration: Pacing Impedance
Description: Subjects' bipolar pacing impedance was measured at implant, pre-hospital discharge and all scheduled follow-up visits. Pacing impedance at the 6 month visit is presented here.
Time Frame: 6 month
Population: Subjects with bipolar configuration pacing impedance at 6 month
Measure: Mean (Standard Deviation); unit: Ohms
Groups:
- Model 4396 LV Lead: Subjects with bipolar configuration pacing impedance at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 135
Ohms | 967.1 (239.2)

22. Secondary Outcome: Characterize Model 4396 Electrical Performance- Bipolar Configuration: Sensing
Description: Bipolar sensing, measured by R-wave amplitude, for the Model 4396 was collected at implant, pre-hospital discharge and all scheduled follow-up visits. Measurements at the 6 month visit are presented here.
Time Frame: 6 month
Population: Subjects with bipolar configuration electrode R-wave amplitude at 6 month.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Model 4396 LV Lead: Subjects with bipolar configuration R-wave amplitude at 6 month.
Arm/Group | Model 4396 LV Lead
Number analyzed (Participants) | 140
mV | 15.0 (7.3)

ADVERSE EVENTS:
Time Frame: Subject enrollment-exit
Description: Reported Adverse Events (AE) were documented on study case report forms as they occurred. Serious AE: AE that led to death, or led to worse health that resulted in: life-threatening illness or injury; a permanent impairment of a body function; hosp.; medical intervention or surgery to prevent permanent impairment to body structure or body function
Arm/Group | Model 4396 LV Lead
Serious Adverse Events (participants affected / at risk) | 76/197
Other Adverse Events (participants affected / at risk) | 27/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model 4396 LV Lead (N=197)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alcoholic withdrawal symptoms (Psychiatric disorders) | 1 (1)
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aneurysm of aortic arch (Cardiac disorders) | 1 (1)
Asystole (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 1 (2)
Bladder cancer (Renal and urinary disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 3 (3)
Central line infection (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chest tenderness (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 1 (2)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 2 (2)
Coronary artery disease aggravated (Cardiac disorders) | 1 (1)
Decompensated heart failure (Cardiac disorders) | 15 (17)
Deep venous thrombosis arm (Vascular disorders) | 1 (1)
Degenerative joint disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Device lead issue (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Effusion pleural (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated pacing threshold (Injury, poisoning and procedural complications) | 3 (3)
Embolism pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolus (Vascular disorders) | 1 (1)
Femoral artery stenosis (Vascular disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fever of unknown origin (General disorders) | 1 (1)
Foot infection (Infections and infestations) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 3 (3)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma (General disorders) | 1 (1)
Herniated disc (Nervous system disorders) | 1 (1)
Hyperkalaemia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Implant site hematoma (General disorders) | 3 (3)
Implant site infection (Infections and infestations) | 1 (1)
Inadequate lead connection (Injury, poisoning and procedural complications) | 1 (1)
Inappropriate phrenic nerve stimulation (Injury, poisoning and procedural complications) | 2 (2)
Insulin hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Intracerebral hemorrhage (Nervous system disorders) | 1 (1)
Laceration of head (Injury, poisoning and procedural complications) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 10 (11)
Loss of capture (Injury, poisoning and procedural complications) | 2 (2)
Loss of control of diabetes (Metabolism and nutrition disorders) | 1 (1)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1)
Multiple organ failure (General disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Near syncope (Nervous system disorders) | 1 (1)
Non ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Prostatic hypertrophy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Spinal column stenosis (Nervous system disorders) | 1 (1)
Sudden cardiac death (Cardiac disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (3)
Transient ischemic attack (TIA) (Nervous system disorders) | 1 (1)
Triple vessel disease (Cardiac disorders) | 1 (1)
Twiddler's syndrome (Injury, poisoning and procedural complications) | 2 (2)
Uncontrolled hypertension (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 10 (10)
Vertigo (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Model 4396 LV Lead (N=197)
Inappropriate phrenic nerve stimulation (Injury, poisoning and procedural complications) | 11 (15)
Inappropriate stimulation of diaphragm (Injury, poisoning and procedural complications) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No